CLINICAL TRIAL: NCT05339581
Title: PILOT Study on the Safety and Efficacy of IMRT Combined With PD-1 Blockade and LEnvatinib as Neoadjuvant TherapY for Hepatocellular Carcinoma With Portal Vein Tumor Thrombus (Vp3) Before Liver Transplantation（iPLENTY-pvtt）
Brief Title: IMRT Plus PD-1 Blockade and Lenvatinib for HCC With PVTT (Vp3) Before Liver Transplantation
Acronym: iPLENTY-pvtt
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: RenJi Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Renji-IIT2022-011
Record Dates: First submitted 2022-04-15; First posted 2022-04-21 (Actual); Last update posted 2022-04-27 (Actual); Status verified 2022-04

CONDITIONS: Liver Cancer; Liver Transplant; Complications; Hepatocellular Carcinoma; Portal Vein Thrombosis; Radiotherapy; Complications
MeSH Terms: conditions — Liver Neoplasms; Carcinoma, Hepatocellular | interventions — Radiotherapy, Intensity-Modulated; pembrolizumab; sintilimab; camrelizumab; tislelizumab; lenvatinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IMRT combined with PD-1 Blockade and Lenvatinib (Experimental): Participants receive PD-1 Blockade (Pembrolizumab，Sintilimab， Camrelizumab，Tislelizumab) 200 mg intravenously on day 1 of a 21-day treatment cycle until >42 days before liver transplantation or unacceptable toxicity develops. Participants receive Lenvatinib Mesylate Capsule (Lenvima®) 8 mg orally once daily until >7 days before liver transplantation.
  Neoadjuvant IMRT will be initiated at the third treatment cycle, and the dose prescription of IMRT is for planning target volume (PTV). The prescription dose to 95%PTV should be ≥50 Gy and ≤60 Gy, and been given in daily dose fractions of 2 Gy, 5 days per week. And the final prescription dose is determined according to dose constraints for organs at risk.
  Interventions: Radiation: intensity-modulated radiotherapy; Combination Product: Pembrolizumab; Drug: Sintilimab; Drug: Camrelizumab; Drug: Tislelizumab; Drug: Lenvatinib Mesylate Capsule
- PD-1 Blockade and Lenvatinib (Active Comparator): Participants receive PD-1 Blockade (Pembrolizumab，Sintilimab， Camrelizumab，Tislelizumab) 200 mg intravenously on day 1 of a 21-day treatment cycle until >42 days before liver transplantation or unacceptable toxicity develops. Participants receive Lenvatinib Mesylate Capsule (Lenvima®) 8 mg orally once daily until >7 days before liver transplantation.
  Interventions: Combination Product: Pembrolizumab; Drug: Sintilimab; Drug: Camrelizumab; Drug: Tislelizumab; Drug: Lenvatinib Mesylate Capsule

INTERVENTIONS:
Radiation: intensity-modulated radiotherapy — Neoadjuvant IMRT will be initiated at the third treatment cycle, and the dose prescription of IMRT is for planning target volume (PTV). The prescription dose to 95%PTV should be ≥50 Gy and ≤60 Gy, and been given in daily dose fractions of 2 Gy, 5 days per week. And the final prescription dose is determined according to dose constraints for organs at risk.
  Other Names: IMRT
  Arms: IMRT combined with PD-1 Blockade and Lenvatinib
Combination Product: Pembrolizumab — Participants receive PD-1 Blockade (Pembrolizumab 200mg，Sintilimab 200mg， Camrelizumab 200mg，Tislelizumab 200mg) 100-200 mg intravenously on day 1 of a regular treatment cycle until >42 days before liver transplantation or unacceptable toxicity develops. Participants receive Lenvatinib Mesylate Capsule (Lenvima®) 8 mg orally once daily until >7 days before liver transplantation.
  Other Names: Keytruda
Drug: Sintilimab — Sintilimab is a recombinant anti-human PD-1 monoclonal antibody.
  Other Names: Tyvyt
Drug: Camrelizumab — Camrelizumab is a humanized anti-human PD-1 monoclonal antibody.
  Other Names: AiRuiKa
Drug: Tislelizumab — Tislelizumab is a recombinant anti-human PD-1 monoclonal antibody.
Drug: Lenvatinib Mesylate Capsule — Lenvatinib (Lenvima®, Eisai China) is a novel angiogenesis inhibitor which targets vascular endothelial growth factor 1-3, fibroblast growth factor receptor 1-4, platelet-derived growth factor receptor β, RET and KIT.
  Other Names: LENVIMA

SUMMARY:
This is a parallel assigned, open-label, perspective trial studying the safety and efficacy of intensity-modulated radiotherapy (IMRT) combined with PD-1 Blockade and Lenvatinib for Hepatocellular Carcinoma (HCC) with Vp3 Portal Vein Tumor Thrombus (PVTT, Japanese Liver Cancer Study Group classification) before liver transplantation.

DETAILED DESCRIPTION:
In most criteria (e.g.Milan, UCSF, Up-to-seven), PVTT remains as an absolute contraindication for liver transplant due to the high rate of recurrence and poor prognosis. Neoadjuvant therapy has induced pathological responses in multiple tumor types and might decrease the risk of postoperative recurrence in HCC. The primary endpoint is the necrosis rate of PVTT and the primary tumor.

Participants receive PD-1 Blockade (Pembrolizumab，Sintilimab， Camrelizumab，Tislelizumab) 200 mg intravenously on day 1 of a regular treatment cycle and Lenvatinib Mesylate Capsule (Lenvima®) 8 mg orally once daily. Neoadjuvant IMRT will be initiated at the third treatment cycle, and the dose prescription of IMRT is for planning target volume (PTV). The prescription dose to 95%PTV should be ≥50 Gy and ≤60 Gy, and been given in daily dose fractions of 2 Gy, 5 days per week. And the final prescription dose is determined according to dose constraints for organs at risk.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have pathologically or cytologically or by radiological criteria proven hepatocellular carcinoma（exceeding Milan criteria）; known mixed histology (e.g. hepatocellular carcinoma plus cholangiocarcinoma) or fibrolamellar variant is not allowed.
* The maximum diameter of a single tumor ≤9cm. Or the number of tumors ≤3 and the maximum diameter of the largest tumors ≤5cm, and the sum of the maximum diameters of all tumors ≤9cm.
* Vp3 PVTT according to Japanese Vp classification.
* Without lymph node metastasis or extrahepatic metastasis.
* Baseline AFP≥20ng/ mL
* Has an eligibility scan (CT of the chest, triphasic CT scan and MRI of the abdomen) <1 week before the treatment.
* Has an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1 within 7 days prior to Cycle 1, Day 1.
* Has a Child-Pugh A-B7 liver score (5 to 7 points) within 7 days prior to Cycle 1, Day 1.
* Laboratory tests within 7 days prior to Cycle 1, Day 1:
* Neutrophils ≥1.5×109/L
* Hemoglobin ≥8.5g/dL
* Platelets ≥100×109/L,
* Creatinine ≤1.5× upper limit of normal (ULN) and endogenous creatinine clearance ≥50ml/min (standard Cockcroft Gaul formula)
* Total bilirubin ≤3×ULN, ALT≤5×ULN, AST≤5×ULN, INR≤1.7
* Has controlled hepatitis B (HBV-DNA<105IU/ml)
* The estimate time length between enrollment and liver transplantation should be at least 3 months.
* No prior systematic therapy such as immunotherapy, targeted therapy and chemotherapy for HCC.
* No prior local treatment such as TACE, HAIC, radiofrequency ablation or radiotherapy was received within 2 months before enrollment.
* If female, is not pregnant or breastfeeding, and at least one of the following conditions applies: 1) Is not a woman of childbearing potential (WOCBP); or 2) Is a WOCBP and using a contraceptive method that is highly effective or be abstinent from heterosexual intercourse as their preferred and usual lifestyle (a WOCBP must have a negative pregnancy test within 72 hours before the first dose of study treatment).
* No obvious insufficiency of other organs.
* Patients with a history of hypertension should be well controlled (< 140/90 mmHg) on a regimen of anti-hypertensive therapy.
* Patients voluntarily joined the study and signed informed consent with good compliance and follow-up.

Exclusion Criteria:

* • Known mixed histology (e.g. hepatocellular carcinoma plus cholangiocarcinoma) or fibrolamellar variant.

  * Surgery within the past 6 months.
  * Has had esophageal or gastric variceal bleeding within the last 6 months.
  * Has clinically apparent ascites on physical examination.
  * Has received systematic therapy such as immunotherapy, targeted therapy and chemotherapy for HCC.
  * Has received TACE, HAIC, radiofrequency ablation and other local treatments in recent 2 months.
  * Has received liver radiotherapy.
  * Has received radiotherapy with grade 4 toxicity.
  * Significant history of cardiac disease is not allowed: Congestive heart failure > class II New York Heart Association (NYHA) Myocardial infarction within 6 months prior to registration Serious myocardial dysfunction, defined as scintigraphically (multigated acquisition scan [MUGA], myocardial scintigram) determined absolute left ventricular ejection fraction (LVEF) below 45% or an LVEF on echocardiogram (ECHO) below the normal limit at the individual institution.
  * Has severe hypersensitivity (≥Grade 3) to monoclonal antibody.
  * Has an active autoimmune disease that has required systemic treatment (skin diseases that do not require systemic treatment such as vitiligo, psoriasis; type I diabetes, and autoimmune hypothyroidism due to hormone replacement therapy are allowed).
  * Patients with other active malignant tumors within 5 years before the first use of the study drug (cured localized tumors such as basal cell carcinoma of skin, squamous cell carcinoma of skin, superficial bladder cancer, carcinoma in situ of prostate, carcinoma in situ of cervix and carcinoma in situ of breast are allowed).
  * Has an active infection requiring systemic therapy.
  * Has a known history of human immunodeficiency virus (HIV) infection.
  * Has known active tuberculosis within 5 years.
  * Has received a live vaccine within 30 days prior to the first dose of study treatment.
  * Has received bone-marrow allotransplantation or solid organ transplantation.
  * Is currently participating in or has participated in a study of an investigational agent or has used an investigational device within 4 weeks prior to Cycle 1, Day 1.
  * Dysphagia or known drug absorption disorder.
  * Is pregnant or breastfeeding or expecting to conceive or father children within the projected duration of the study, starting with the screening visit through 120 days after the last dose of study treatment.
  * Conditions considered unsuitable for inclusion by other researchers.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Estimated)
Dates: Start 2022-05-20 (Estimated); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-05-31 (Estimated)

PRIMARY OUTCOMES:
PVTT RR/NR | up to 12 months
  Portal vein tumor thrombus related Response and Necrosis Rate

SECONDARY OUTCOMES:
Alpha Fetoprotein Response (AFP-R) | up to 12 months
  AFP-R is defined as a >20% decrease in AFP serum level from baseline to the time of liver transplant, if liver transplant is not possible, the final AFP level would be measured as the AFP level at 12 months.
Progression-free survival (PFS) | up to 12 months
  PFS is defined as the time from the date of treatment initiation to the date of the first observation of progressive disease (PD) by independent radiologic review according to mRECIST criteria or death from any cause.
Objective Response Rate (ORR) | up to 12 months
  RR is defined as the proportion of patients whose tumor volume has reached a predetermined value and can maintain a minimum time limit, including complete response(CR) and partial response(PR) by independent radiologic review according to mRECIST criteria.
Time to Progression (TTP) | up to 12 months
  TTP is defined as the duration from the date of patient recruited to the first progress at any site or the date of death from any cause.
Duration of response (DOR) | up to 12 months
  DOR is defined as the duration from the date that measurement criteria are met for CR or PR to the first progress at any site or the date of death from any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Qiang Xia, MD, Ph.D, Study Chair — Dept. Liver Surgery, Renji Hospital, School of Medicine, SJTU; Yong-rui Bai, MD, Study Chair — Dept. Radiotherapy, Renji Hospital, School of Medicine, SJTU; Xiu-mei Ma, MD, Principal Investigator — Dept. Radiotherapy, Renji Hospital, School of Medicine, SJTU; Xiao-hang Wang, MD, Principal Investigator — Dept. Radiotherapy, Renji Hospital, School of Medicine, SJTU; Hao Feng, MD, Ph.D, Principal Investigator — Dept. Liver Surgery, Renji Hospital, School of Medicine, SJTU
Locations (1):
- Ren Ji Hospital, School of Medicine, Shanghai Jiao Tong University, Shanghai, China